CLINICAL TRIAL: NCT05733182
Title: Effect of Colour Temperature of Reading Lamp on Refractive Error Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr CHOI Kai Yip, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00000
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Refractive Errors
Keywords: Myopia; Environment; Colour temperature; Lighting
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3000K (Active Comparator): Participants will receive a reading lamp of colour temperature 3000K.
  Interventions: Device: 3000K Reading lamp
- 4500K (Active Comparator): Participants will receive a reading lamp of colour temperature 4500K.
  Interventions: Device: 4500K Reading lamp
- 6500K (Active Comparator): Participants will receive a reading lamp of colour temperature 6500K.
  Interventions: Device: 6500K Reading lamp

INTERVENTIONS:
Device: 3000K Reading lamp — Reading lamp with custom-made circuitry to emit light of 3000K colour temperature
  Arms: 3000K
Device: 4500K Reading lamp — Reading lamp with custom-made circuitry to emit light of 4500K colour temperature
  Arms: 4500K
Device: 6500K Reading lamp — Reading lamp with custom-made circuitry to emit light of 6500K colour temperature
  Arms: 6500K

SUMMARY:
This is a 12-month longitudinal randomized controlled trial aiming to evaluate the effect of colour temperature of reading lamp on refractive error development.

DETAILED DESCRIPTION:
Myopia has reached epidemic in the world, especially in East Asia. The proportion of myopic population increases drastically during schoolage. Lack of light exposure has been suggested to be a risk for myopia development, in which additional reading lamp may alleviate this condition. However, the effect of colour temperature of the reading lamp is unknown on childhood refractive error development. In this study, investigators will randomly allocate school-aged children into groups, who will receive reading lamps of different colour temperatures for their daily use. The participants' refractive error and axial length will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged between 4 and 18 years

Exclusion Criteria:

* have received myopia control intervention

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 798 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refraction | up to 12 months
  Refractive error in diopter by autorefractor
Axial length | up to 12 months
  Length of the eyeball in millimeter by partial coherence interferometer

SECONDARY OUTCOMES:
Colour vision | up to 12 months
  Ability to distinguish colours (pass/fail & severity of defect) measured by pseudoisochromatic plates

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Research Clinic, Hong Kong, Kowloon, Hong Kong